CLINICAL TRIAL: NCT00002008
Title: An Open Label Phase I Study of Subcutaneously Administered Recombinant Human GM-CSF in Patients With AIDS Virus Infection and Leukopenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 067D; 106
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-01

CONDITIONS: HIV Infections; Cytopenias
Keywords: Leukopenia; Drug Evaluation; Granulocyte-Macrophage Colony-Stimulating Factor
MeSH Terms: conditions — HIV Infections; Cytopenia; Leukopenia | interventions — sargramostim

INTERVENTIONS:
Drug: Sargramostim

SUMMARY:
To determine the safety, immunogenicity, biological activity, ad pharmacokinetics of sargramostim ( recombinant granulocyte-macrophage colony-stimulating factor; GM-CSF ) human granulocyte-macrophage colony-stimulating factor ( GM-CSF ), given by subcutaneous ( SC ) injection to patients with leukopenia in association with HIV infection.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Serum antibody to HIV with or without evidence of HIV.
* Antigenemia.
* Anticipated survival of at least 6 months.
* Allowed:
* Kaposi's sarcoma.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Malignancy other than Kaposi's sarcoma.
* Excessive diarrhea (more than 5 liquid or non-liquid stools per day).
* Currently hospitalized or hospitalized within the last 4 weeks for the treatment of opportunistic infection.
* Primary hematologic or infectious disorders unrelated to AIDS virus infection.
* Dementia or altered mental status that would prohibit the giving and understanding of informed consent.

Patients with the following are excluded:

* History of malignancy other than Kaposi's sarcoma.
* Currently hospitalized or hospitalized within 4 weeks for the treatment of opportunistic infection.

Prior Medication:

Excluded within 3 weeks of study entry:

* Marrow suppressive medication.
* Excluded within 4 weeks of study entry:
* Any investigational drug.

Prior Treatment:

Excluded within 4 weeks of study entry:

* Systemic cytotoxic chemotherapy.
* Irradiation.

Risk Behavior:

Excluded within 3 months of study entry:

* Regular, excessive users of alcohol, hallucinogens, or agents which are addicting.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA CARE Ctr, Los Angeles, California
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts